CLINICAL TRIAL: NCT00682188
Title: A School Nurse-Delivered Intervention for Overweight and At Risk Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Lori Pbert, Professor of Medicine, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21HD053371 (NIH)
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Adolescents; Youth; School health; Randomized controlled trial; Intervention study
MeSH Terms: conditions — Overweight; Obesity | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CI (Experimental): Six 30-minute individual student-centered counseling sessions based on the 5A approach to assist adolescents in making changes in their diet and level of physical activity delivered by school nurses over 2 months (weekly in month 1, biweekly in month 2)
  Interventions: Behavioral: Counseling Intervention
- II (Active Comparator): Six individual sessions with the school nurse over 2 months to check weight and behavior changes and provide a series of six pamphlets on weight and weight management
  Interventions: Behavioral: Information Intervention

INTERVENTIONS:
Behavioral: Counseling Intervention — Six 30-minute individual student-centered counseling sessions based on the 5A approach to assist adolescents in making changes in their diet and level of physical activity delivered by school nurses over 2 months (weekly in month 1, biweekly in month 2)
  Arms: CI
Behavioral: Information Intervention — Six individual sessions with the school nurse over 2 months to check weight and behavioral changes and provide a series of six pamphlets on weight and weight management
  Arms: II

SUMMARY:
Overweight in adolescents has nearly tripled in the past two decades and has serious physical and psychosocial consequences, both during adolescence and into adulthood. School nurses have tremendous potential to prevent and treat overweight in this population, as over 95% of adolescents have contact with the school health system each year and school nurses have the credibility and skills to provide guidance regarding weight, diet and physical activity. The goals of the proposed exploratory study are to adapt an innovative, theory-based school nurse-delivered counseling intervention model used effectively for smoking cessation for the treatment of adolescent overweight, and test its feasibility and potential efficacy in reducing BMI, improving diet, increasing physical activity and decreasing sedentary behavior. If the results of this exploratory study prove promising, the efficacy of the intervention will be evaluated in a large scale randomized controlled trial.

DETAILED DESCRIPTION:
Overweight in adolescents has nearly tripled in the past two decades and has serious physical and psychosocial consequences, both during adolescence and into adulthood. School nurses have tremendous potential to identify, prevent, and treat overweight in this population, as over 95% of children and adolescents have contact with the school health system each year and school nurses have the credibility and skills to provide guidance regarding weight, diet and physical activity. However, to our knowledge there have been no randomized controlled school-based trials that have utilized the school nurse to deliver weight-related intervention to adolescents. In a RCT conducted by the investigators, we found a school nurse-delivered smoking cessation intervention was successful in assisting adolescent smokers to quit, being both feasible to deliver in the school health setting and very well received by adolescents.

This two-year exploratory study will adapt this innovative, theory-based school nurse-delivered intervention model for the treatment of adolescent overweight, and test its feasibility and potential efficacy in reducing BMI, improving diet, increasing physical activity and decreasing sedentary behavior. The content of the intervention will be based on current clinical guidelines for the treatment of overweight in adolescents and Social Cognitive Theory (SCT), employing cognitive-behavioral techniques to facilitate changes in a set of very focused self-management behaviors: diet (at least 5 fruits vegetables a day; avoid soda and sugar sweetened drinks), physical activity (at least 1 hour on most days), and sedentary behavior (less than 2 hours of TV, video, and computer time a day). Four high schools in Massachusetts will be pair matched on demographics, school size, and percent low income and randomly assigned to one of two conditions: (1) Counseling Intervention (CI) consisting of six 30-minute individual student-centered counseling sessions delivered by school nurses over 2 months (weekly in month 1, biweekly in month 2); or (2) Information Intervention (II) attention-control comparison condition consisting of six individual sessions with the school nurse over 2 months (weekly in month 1, biweekly in month 2) to check status regarding weight and behavior changes and deliver a series of standardized pamphlets on weight and weight management. Adolescents (n=84) enrolled in grades 9 through 12 at-risk for overweight (body mass index (BMI) between the 85th and 94th percentile for age and gender) or overweight (BMI at or greater than the 95th percentile) will be recruited from the four schools. Assessments will be conducted at baseline and at 3-and 6-month follow-up. Should the results of this exploratory study prove promising the efficacy of the intervention will be evaluated in a large scale RCT. If found to be effective, such a school nurse-delivered intervention for adolescent overweight would have tremendous potential for wide-scale dissemination.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in grades 9 through 12
* BMI equal or greater than 85th percentile
* able to understand and participate in study protocol
* able to provide informed assent (adolescent) and consent (parent)
* student and at least one parent English speaking

Exclusion Criteria:

* unable/unwilling to provide informed assent (adolescent)and consent (parent)
* planning to move out of the area within the next 6 months
* medical condition that precludes adherence to study dietary recommendations
* diagnosis of a serious psychiatric illness within the past 5 years
* genetic or endocrine causes of obesity
* developmental delay that would prevent participation in intervention or measurements
* prescribed medications associated with weight gain
* morbidly obese, defined as 300 pounds oe greater

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2008-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
BMI | 3- and 6-month post baseline

SECONDARY OUTCOMES:
Adherence to self-management behaviors (diet, physical activity, and sedentary behavior) | 3- and 6-month post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Lori Pbert, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States